CLINICAL TRIAL: NCT01974089
Title: Oropharyngeal Dysphagia in Patients With Community Acquired Pneumonia
Status: Completed | Type: Observational
Sponsor: Regionshospital Nordjylland (Other Government)
Responsible Party: Principal Investigator, Dorte Melgaard Kristiansen, Developmental therapist, phd, Regionshospital Nordjylland
Other Study IDs: RHN_DMK_03
Record Dates: First submitted 2013-10-25; First posted 2013-11-01 (Estimated); Results first posted 2018-10-01 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Dysphagia; Pneumonia
Keywords: Dysphagia; Community acquired pneumonia; Mortality; Rehospitalization
MeSH Terms: conditions — Deglutition Disorders; Pneumonia; Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pneumonia and dysphagia: Patients with community aquired pneumonia and oropharyngea dysphagia
  Interventions: Other: Dysphagia
- Pneumonia: Patients with community aquired pneumonia

INTERVENTIONS:
Other: Dysphagia — Oropharyngeal dysphagia assessed by Volume-Viscosity Svallowing Test
  Groups: Pneumonia and dysphagia

SUMMARY:
This study investigates relationship between community acquired pneumonia and oropharyngeal dysphagia in patients admitted to a department of respiratory medicine in Northern Denmark.

The endpoints will be re-hospitalisation and mortality.

DETAILED DESCRIPTION:
Community acquired pneumonia (CAP) is an important cause of morbidity and mortality in elderly patients. Risk factors are many including oropharyngeal dysphagia (OD). Systematic screening of OD is recommended for at-risk popolations, however these resommandations do not specifically address elderly patients hospitalized with CAP.

In this study OD is assessed in all patients by Volume-Viscosity Swallowing Test (V-VST) The study is registered by the Danish Data Protection Authority (2008-58-0028)

ELIGIBILITY:
Inclusion Criteria:

* Temperature > 38 degrees Celcius
* New infiltrate on chest x-ray
* Increased C-reactive protein (CRP)
* Either cough, dyspnea, pleuritic chest pain, expectoration, or tachypnea

Exclusion Criteria:

* patients referred from the intensive care unit
* reduced cognitive awareness if not able to able to cooperate with the assessment of oropharyngeal dysphagia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients recruited from the Department of Respiratory Medicine at North Denmeark Regional Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2013-10; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vendsyssel Hospital, Hjørring, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- Pneumonia and Dysphagia: Patients with community acquired pneumonia and oropharyngeal dysphagia
- Pneumonia: Patients with community acquired pneumonia
Period: Overall Study
Arm/Group | Pneumonia and Dysphagia | Pneumonia
Started | 53 | 101
Completed | 53 | 101
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pneumonia and Dysphagia | Pneumonia | Total
Number analyzed (Participants) | 53 | 101 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 23 | 30
  >=65 years | 46 | 78 | 124
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 50 | 70
  Male | 33 | 51 | 84
Region of Enrollment [Number; unit: participants]
  Denmark | 53 | 101 | 154

OUTCOME MEASURES:

1. Primary Outcome: Intra Hospital Mortality
Description: Intra hospital mortality is death while the patient is hospitalized
Time Frame: With in 10 days from admission
Measure: Count of Participants; unit: Participants
Arm/Group | Pneumonia and Dysphagia | Pneumonia
Number analyzed (Participants) | 53 | 101
Participants | 7 | 0

2. Primary Outcome: 30 Day Mortality
Description: Death within 30 days of discharge
Time Frame: 30 days after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Pneumonia and Dysphagia | Pneumonia
Number analyzed (Participants) | 46 | 101
Participants | 10 | 2

3. Primary Outcome: Re-hospitalization
Description: The rate of re-hospitalization within 30 days of discharge
Time Frame: 30 days after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Pneumonia and Dysphagia | Pneumonia
Number analyzed (Participants) | 46 | 101
Participants | 10 | 15

ADVERSE EVENTS:
Time Frame: Adverse events reported until 30 days after discharge from hospital
Arm/Group | Pneumonia and Dysphagia | Pneumonia
All-Cause Mortality (participants affected / at risk) | 17/53 | 2/101
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/101
Other Adverse Events (participants affected / at risk) | 0/53 | 0/101

LIMITATIONS AND CAVEATS:
Small sample size. The definition of community acquired pneumonia is vague and unclear and there is a risk that some patients may be hospitalized with aspiration pneumonia, a subtype of community acquired pneumonia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes